CLINICAL TRIAL: NCT00952484
Title: A Randomized, Open-Label, Multicenter, Multinational, Dose-Ranging, Historical Control Study of the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of ENB-0040 (Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein) in Children With Hypophosphatasia (HPP)
Brief Title: Safety and Efficacy of Asfotase Alfa in Juvenile Patients With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENB-006-09
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 mg/kg (Active Comparator): 2 mg/kg subcutaneous injection three times per week.
  Interventions: Biological: asfotase alfa
- 3 mg/kg (Active Comparator): 3 mg/kg subcutaneous injection three times per week.
  Interventions: Biological: asfotase alfa

INTERVENTIONS:
Biological: asfotase alfa — 2 mg/kg subcutaneous injection three times per week for 6 months.
  Other Names: Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein; sALP-Fc-D10
  Arms: 2 mg/kg
Biological: asfotase alfa — 3 mg/kg subcutaneous injection three times per week for 6 months.
  Other Names: Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein; sALP-Fc-D10
  Arms: 3 mg/kg

SUMMARY:
This clinical trial studied the safety and efficacy of asfotase alfa in children with HPP compared to a historical control group.

DETAILED DESCRIPTION:
Asfotase Alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

Efficacy analyses were prospectively defined in the protocol with a comparison to historical controls. The historical control group came from patients whose characteristics matched as closely as possible the entry criteria for the trial. The control group included all patients who had x-rays within the age range defined by the inclusion criteria of this study (5 to 12 years of age, inclusive, with open growth plates).

The pre-specified plan for analysis was to combine the two asfotase alfa treated groups (asfotase alfa 2 mg/kg subcutaneous (SC) injection three times per week or 3 mg/kg subcutaneous (SC) injection three times per week) and compare them to historical controls.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from parent or legal guardian prior to participation
2. Patients > 5 and < 12 years of age with open growth plates at time of enrollment
3. Tanner stage of 2 or less indicating pre-pubescence
4. Documented history of HPP, as evidenced by:

   * Presence of HPP-related rickets on skeletal radiographs of the wrist and knee
   * Serum alkaline phosphatase (ALP) below age-adjusted normal range
   * Plasma PLP at least twice the upper limit of normal
5. 25(OH) vitamin D level > 20 ng/mL
6. Ability of patient and parent/guardian to comply with study requirements

Exclusion Criteria:

1. Serum calcium or phosphorus below age-adjusted normal range
2. History of sensitivity to any study drug constituent
3. Medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities
4. Treatment with an investigational drug within 1 month before start of study drug
5. Current enrollment in any other study involving an investigational new drug, device, or treatment for HPP (e.g., bone marrow transplantation)
6. Current evidence of a treatable form of rickets
7. Prior treatment with bisphosphonates
8. Bone fracture or orthopedic surgery within the past 12 months that, in the opinion of the Investigator would interfere with the ability of study patient to comply with study protocol
9. Major congenital abnormality other than those associated with HPP

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Shriners Hospital for Children, St Louis, Missouri, United States
- The University of Manitoba Health Services Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Millan JL, Narisawa S, Lemire I, Loisel TP, Boileau G, Leonard P, Gramatikova S, Terkeltaub R, Camacho NP, McKee MD, Crine P, Whyte MP. Enzyme replacement therapy for murine hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):777-87. doi: 10.1359/jbmr.071213. PMID 18086009
- [Derived] Simmons JH, Rush ET, Petryk A, Zhou S, Martos-Moreno GA. Dual X-ray absorptiometry has limited utility in detecting bone pathology in children with hypophosphatasia: A pooled post hoc analysis of asfotase alfa clinical trial data. Bone. 2020 Aug;137:115413. doi: 10.1016/j.bone.2020.115413. Epub 2020 May 14. PMID 32417537
- [Derived] Whyte MP, Madson KL, Phillips D, Reeves AL, McAlister WH, Yakimoski A, Mack KE, Hamilton K, Kagan K, Fujita KP, Thompson DD, Moseley S, Odrljin T, Rockman-Greenberg C. Asfotase alfa therapy for children with hypophosphatasia. JCI Insight. 2016 Jun 16;1(9):e85971. doi: 10.1172/jci.insight.85971. PMID 27699270
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited to participate in the study from September to December 2009 at investigational sites via posting in clinicaltrials.gov and contact with physicians experienced in the diagnosis and management of HPP. De-identified historical controls were also selected from a natural history database of patients with HPP.
Pre-assignment Details: Patients meeting eligibility criteria were randomly assigned to receive 2mg/kg or 3mg/kg of asfotase alfa SC 3 times weekly for 24 weeks.
Groups:
- 2 mg/kg Asfotase Alfa: 2 mg/kg subcutaneous (SC) injection three times per week.
- 3 mg/kg Asfotase Alfa: 3 mg/kg subcutaneous (SC) injection three times per week.
- Historical Control: De-identified historical control patients (i.e., untreated with asfotase alfa) were selected from a longitudinal natural history database of patients with HPP maintained at Shriner's Hospitals for Children, St. Louis, Missouri.
  Historical controls must have had at least two sets of wrist and knee radiographs taken between the ages of 5 years, 0 months and 12 years, 0 months with evidence of open growth plates.
Period: Overall Study
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa | Historical Control
Started | 6 | 7 | 16
Completed | 6 | 6 | 16
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asfotase Alfa 2 mg/kg: 2 mg/kg thrice weekly administered as a subcutaneous (SC) injection
- Asfotase Alfa 3 mg/kg: 3 mg/kg administered thrice weekly as a subcutaneous (SC) injection
- Historical Control: De-identified historical controls selected from a natural history database of patients with HPP.
- Total: Total of all reporting groups
Arm/Group | Asfotase Alfa 2 mg/kg | Asfotase Alfa 3 mg/kg | Historical Control | Total
Number analyzed (Participants) | 6 | 7 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 16 | 29
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (2.2) | 9.1 (2.3) | 6.0 (1.78) | 7.3 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 5 | 7
  Male | 5 | 6 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 16 | 25
  Canada | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Rickets Severity on Skeletal Radiographs From Baseline to Week 24 as Measured by the Radiographic Global Impression of Change (RGI-C) Scale
Description: A 7-point RGI-C (radiographic global impression of change) score was used to rate change in rickets severity. Only those patients with a minimum score of +2 indicating substantial healing of rickets) were considered responders. Three pediatric radiologists not affiliated with the conduct of the study performed the ratings.
Time Frame: Baseline and Week 24
Population: ITT population, which included randomized patients that received treatment with asfotase alfa, even if discontinued or lost to follow-up. The last assessment prior to Week 24 is used for missing Week 24 data; patients with no post-baseline assessments imputed as having no change. A historical control group is used for comparison.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Historical Controls: De-identified historical controls selected from a natural history database of patients with HPP.
- Asfotase Alfa Combined: ITT Population: Asfotase alfa 2 mg/kg subcutaneous (SC) injection three times per week or 3 mg/kg subcutaneous (SC) injection three times per week.
Arm/Group | Historical Controls | Asfotase Alfa Combined
Number analyzed (Participants) | 16 | 13
units on a scale | 0 [-1.3 to 2.0] | 2.00 [0.0 to 2.3]
Statistical Analysis 1: Comparison: Historical Controls vs Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.0007, Wilcoxon (Mann-Whitney) — P-value based on Wilcoxon rank sum test comparing the median RGI-C score for the asfotase alfa combined reporting group to the historical control group

2. Secondary Outcome: Change in Osteomalacia - Osteoid Thickness (as Measured by Trans-iliac Crest Bone Biopsy)
Description: Change from Baseline to Week 24 in osteoid thickness.
Time Frame: Baseline and Week 24
Population: ITT population, which included all randomized patients that received any treatment with asfotase alfa (2 mg/kg or 3 mg/kg thrice weekly), even if they discontinued or were lost to follow-up during the conduct of the clinical trial. Data imputation was not performed.
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
um | -3.858 (4.2784)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.0097, t-test, 2 sided — P-value testing whether the mean change from Baseline differs from Zero based on a t-test

3. Secondary Outcome: Change in Osteomalacia - Osteoid Volume/Bone Volume (as Measured by Trans-iliac Crest Bone Biopsy)
Description: Change from Baseline to Week 24 in osteoid volume/bone volume (%), calculated as the absolute difference of the Baseline and Week 24 percentages.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
percentage points | -4.225 (7.5582)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.0789, t-test, 2 sided — P-value testing whether the mean change from Baseline differs from Zero based on a t-test

4. Secondary Outcome: Change in Osteomalacia - Mineralization Lag Time (as Measured by Trans-iliac Crest Bone Biopsy)
Description: Change from Baseline to Week 24 in mineralization lag time.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
days | 20.392 (208.9814)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.7417, t-test, 2 sided — P-value testing whether the mean change from Baseline differs from Zero based on a t-test

5. Secondary Outcome: Change in Height (Z-scores)
Description: Change from Baseline to Week 24 in Height Z-Score. Height Z-Scores assigned based on Centers for Disease Control (CDC) growth charts and methodology.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Height Z score
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
Height Z score | 0.01 (0.141)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.7570, Wilcoxon Signed-Rank — P-value testing whether the mean change from Baseline differs from Zero based on a Wilcoxon Signed-Rank test

6. Secondary Outcome: Change in Biomarkers of Asfotase Alfa Activity as Measured by Plasma Inorganic Pyrophosphate (PPi)
Description: Change from Baseline to Week 24 in Plasma PPi
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
uM | -1.883 (0.7285)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value testing whether the mean change from Baseline differs from Zero based on a t-test

7. Secondary Outcome: Change in Biomarkers of Asfotase Alfa Activity as Measured by Pyridoxal-5'-Phosphate (PLP)
Description: Change from Baseline to Week 24 in Plasma PLP
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Asfotase Alfa Combined
Number analyzed (Participants) | 12
ng/mL | -164.533 (121.4840)
Statistical Analysis 1: Comparison: Asfotase Alfa Combined; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided — P-value testing whether the mean change from Baseline differs from Zero based on a t-test

8. Secondary Outcome: Maximum Serum Concentration of Asfotase Alfa (Cmax).
Description: Maximum serum concentration observed following single dose of asfotase alfa.
Time Frame: Study Week 1 (0 to 48 hours post-dose)
Population: ITT population which included all randomized patients that received any treatment with asfotase alfa (2 mg/kg or 3 mg/kg thrice weekly).
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
U/L | 566 (120) | 1260 (439)

9. Secondary Outcome: Time at Maximum Serum Concentration of Asfotase Alfa (Tmax)
Description: Maximum serum concentration observed following single dose of asfotase alfa.
Time Frame: Study Week 1 (0 to 48 hours post-dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
hours | 37.2 (8.1) | 34.3 (6.0)

10. Secondary Outcome: Area Under Serum Concentration-time Curve to Last Measurable Concentration of Asfotase Alfa (AUCt)
Description: Area under serum concentration-time curve to last measurable concentration following single dose of asfotase alfa.
Time Frame: Study Week 1 (0 to 48 hours post-dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*U/L
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
h*U/L | 19700 (5720) | 45200 (15100)

11. Secondary Outcome: Maximum Serum Concentration of Asfotase Alfa (Cmax).
Description: Maximum serum concentration observed following multiple doses of asfotase alfa.
Time Frame: Study Week 6 (0 to 48 hours post-dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
U/L | 1780 (666) | 2280 (875)

12. Secondary Outcome: Time at Maximum Serum Concentration of Asfotase Alfa (Tmax).
Description: Time at maximum serum concentration observed following multiple doses of asfotase alfa.
Time Frame: Study Week 6 (0 to 48 hours post-dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
hours | 20.8 (10) | 17.3 (8.6)

13. Secondary Outcome: Area Under Serum Concentration-time Curve to Last Measurable Concentration of Asfotase Alfa (AUCt)
Description: Area under serum concentration-time curve to last measurable concentration following multiple doses of asfotase alfa.
Time Frame: Study Week 6 (0 to 48 hours post-dose).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*U/L
Arm/Group | 2 mg/kg Asfotase Alfa | 3 mg/kg Asfotase Alfa
Number analyzed (Participants) | 6 | 7
h*U/L | 76000 (28100) | 94200 (44400)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event data for the historical control group were not collected.
Arm/Group | Asfotase Alfa 2 mg/kg | Asfotase Alfa 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa 2 mg/kg (N=6) | Asfotase Alfa 3 mg/kg (N=7)
Injection site erythema (General disorders) | 5 (13) | 7 (16)
Injection site discoloration (General disorders) | 4 (4) | 4 (4)
Injection site pruritis (General disorders) | 4 (8) | 3 (3)
Injection site pain (General disorders) | 3 (5) | 3 (5)
Injection site swelling (General disorders) | 1 (3) | 2 (2)
Infusion site pain (General disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (8) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Blood 1,25-dihydroxycholecaliferol decreased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 1 (1)
Scleral hemmorhage (Eye disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eye Allergy (Eye disorders) | 1 (1) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site hemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Edema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 1 (1) | 0 (0)
Vitamin B6 decreased (Investigations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less